CLINICAL TRIAL: NCT03377010
Title: UF-BMT-HSCT-001: A Non-Interventional Study Evaluating the Quality of Diet in Allogeneic and Autologous Hematopoietic Stem Cell Transplant Survivors
Brief Title: UF-BMT-HSCT-001: A Non-Interventional Study Evaluating Diet in HSCT Survivors
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201702189; UF-BMT-HSCT-001 (Other: University of Florida); OCR16001 (Other: Universiy of Florida)
Record Dates: First submitted 2017-12-13; First posted 2017-12-19 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Hematopoietic Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hematopoietic Stem Cell Transplant (HSCT) Survivor: Study participants will be administered a Dietary Intake - Food Frequency Questionnaire and a Receptivity to Participating in Diet Interventions Questionnaire.
  Interventions: Other: Dietary intake -Food Frequency Questionnaire; Other: Receptivity to Participating in Diet Interventions

INTERVENTIONS:
Other: Dietary intake -Food Frequency Questionnaire — Dietary intake will be assessed using 2014 full-length food frequency questionnaire. The Block 2014 questionnaire combines a full-length food frequency questionnaire with a brief physical activity screening tool. The food and beverage list includes 127 items in the past 1 month, plus additional questions to adjust for fat, protein, carbohydrate, sugar, and whole grain content.
Other: Receptivity to Participating in Diet Interventions — Study participants will rate their interest in learning more about dietary interventions to stay healthy using items developed specifically for this study. The items will be rated on a 3-point Likert-type scale from 3 (extremely interested) to 1 (not at all interested).

SUMMARY:
This is a single center, cross-sectional, non-interventional study aimed at the nutritional intake of long-term health of allogeneic or autologous hematopoietic stem cell transplant (HSCT) survivors.

DETAILED DESCRIPTION:
Higher rates of comorbidity among hematopoietic stem cell transplant (HSCT) survivors support the need for lifestyle interventions that target this vulnerable population. Comprehensive evaluation of the nutrient intake will provide adequate information necessary for develop of a targeted nutritional intervention in order to achieve specific nutritional need and improve long-term health of HSCT survivors. The cross-sectional design of this study has been selected for the timely collection of subject reported nutrient intake data. The intended study is strictly observational.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject and the ability for the subject to comply with all the study-related procedures for subjects enrolled from the cancer registry.
* Both males and females ≥ 18 years of age.
* A medical history of allogeneic or autologous hematopoietic stem cell transplant (HSCT), irrespective of the disease. For the purpose of this study, HSCT survivor is defined as subjects one or more years after allogeneic or autologous HSCT without disease relapse, active graft-versus-host disease, or active infection. Subjects with chronic graft versus host disease who are on stable dose of immunosuppressant (or being tapered off of immunosuppressant) over the past 3 months will be eligible.
* Study participants must have the ability to complete the questionnaires through one of the previously stated mechanisms.
* English speaking due to the logistics of the questionnaires and phone contact included in this study.

Exclusion Criteria:

* Subjects demonstrating an inability to comply with the study procedures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both males and females who have a medical history of allogeneic or autologous hematopoietic stem cell transplant (HSCT), irrespective of the disease. For the purpose of this study, HSCT survivor is defined as subjects one or more years after allogeneic or autologous HSCT without disease relapse, active graft-versus-host disease, or active infection.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2017-12-14 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
Diet intake | 1 month
  To evaluate the diet intake of long-term survivors of HSCT

CONTACTS AND LOCATIONS:
Overall Officials: Nosha Farhadfar, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Cancer Center, Gainesville, Florida, United States